## e-Natureza: Affective Validation of Nature Images as a Complementary Resource for Promoting Well-being in Hospital Environment

## INFORMED CONSENT FORM

Sao Paulo, Brazil

Approved in the first version in 01/31/2017

Human subjects protection review board number: Hospital Israelita Albert Einstein Research Ethics Committee 64096816.9.0000.0071.

## INFORMED CONSENT FORM

Patient

Principal researcher: Eliseth Ribeiro Leão

Research title: "E-NATUREZA: AFFECTIVE VALIDATION OF NATURE IMAGES AS A COMPLEMENTARY RESOURCE FOR PROMOTING WELL-

BEING IN HOSPITAL ENVIRONMENT"

| Name (participant): |
|---------------------|
| Dear participant. |

We would like to invite you to participate as a research volunteer entitled "E-NATUREZA: AFFECTIVE VALIDATION OF NATURE IMAGES AS A COMPLEMENTARY RESOURCE FOR PROMOTING WELL-BEING IN HOSPITAL ENVIRONMENT". The objective of this study is to identify if nature photographs may have some influence on you while you are receiving chemotherapy treatment.

INVOLVEMENT IN THE RESEARCH: By participating in this study you commit to watch a video with nature pictures and then answer some questionnaires to measure the symptoms during the chemotherapy, as well as your state of mind. You will also fill out some data such as age, schooling so that we can characterize the participants in this research.

Because this is a clinical trial, you can be in the intervention group or in the control group. If you join the control group, you will only have to respond the questionnaires, but you will not see the video. If you are interested, after you have answered the questionnaires, we can show the video to you.

We remind you that your participation is voluntary and you have freedom to refuse participating and may still stop responding at any time without any prejudice. In addition, you still have the right to keep one of the copies of the consent form. Whenever you want you can ask more information about the research. To do this, you can contact the researcher, by the means informed below, in this document.

RISK AND DISCOMFORT: The participation in this research presents minimum risks, perhaps only, some embarrassment (shame) that some people feel when they are providing information about themselves.

RESEARCH CONFIDENTIALITY: All information collected in this study are

strictly confidential. Your name will not be mentioned in any moment. All data

will be analyzed together, ensuring the anonymity of the information. The results

may be used in events and scientific publications.

BENEFITS: If you are drawn to the intervention group maybe the video will

bring some sense of well-being for you during your chemotherapy session, but

we do not know, so we are doing this study. If you are drawn for the control

group we do not expect immediate and direct benefits for you for your

participation, but the results will contribute to a new form of intervention that

benefits patients in hospitals if show effective.

PAYMENT: You will not have any expenses for participating in this research.

And nothing will be paid for your participation. However, if you want, you may

have access to copies of the research reports containing the results of this

study. To do so, you just have to contact the responsible researcher as follows:

Address of the person in charge of the research:

Name: Eliseth Ribeiro Leão

Institution: Instituto Israelita de Ensino e Pesquisa

Address: Av. Albert Einstein 627/700 - Block A - 2nd floor

Contact Phones: (55 11) 2151- 1032

CAUTION: To report irregular occurrences or to obtain information on the

ethical aspects of the study, during their participation, please contact:

Research Ethics Committee of the Hospital Israelita Albert Einstein

Av. Albert Einstein, 627/700 - Block A, 2°ss

Morumbi - São Paulo - SP- 05652-000

Tel.: (55 11) 2151-3729

Fax.: (55 11) 2151-0273

PARTICIPATION CONSENT AS A PARTICIPANT

3

I understand that I am free to accept or refuse to participate and that I can with draw my authorization and leave the study at any time. By signing this Informed Consent Form, I am not relinquishing my legal rights. I will receive a signed and dated copy of this Informed Consent Form.

Having fully understood of everything that was told me about my participation in the mentioned study and being aware of my rights, my responsibilities, the risks and the benefits that my participation implies, I agree to participate in it and for this I EXPRESS MY CONSENT WITHOUT FOR THAT I HAVE BEEN FORCED OR OBLIGED.

We thank you for your attention and participation and we make ourselves available for more information about the study at any time.

| Date:// | |
|---|---|
| Participant's Name and Signature | - ———————————————————————————————————— |
| Name and Signature of the researcher applying t | the Term |